CLINICAL TRIAL: NCT06896799
Title: Determining the Effect of Food Ordering on Blood Glucose In Gestational Diabetes Mellitus (DEFI-GDM) - a Randomised Crossover Study
Brief Title: Determining the Effect of Food Ordering on Blood Glucose In Gestational Diabetes Mellitus (DEFI-GDM)
Acronym: DEFI-GDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 25/NI/0004
Record Dates: First submitted 2025-03-04; First posted 2025-03-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational Diabetes Mellitus; Post-prandial glycaemia; Food Ordering
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: This will be a randomised crossover study. Participants will be asked to eat either the protein/fat-based component of the meal (scrambled egg) before or after the carbohydrate-based component (wholemeal toast) on their first visit and on the other visit they will be asked to eat the meal in the reverse order. The order in which this occurs will be randomised and each participant will act as their own control.
Masking Description: It is not possible to blind participants or researchers in this study due to the nature of the nutritional intervention. However, the allocation to each group will be blinded using envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visit 1: Protein/fat then carbohydrate. Visit 2: Carbohydrate then protein/fat. (Experimental): Participants who are randomised to eat the protein/fat-based component (scrambled egg) of the meal before the carbohydrate-based component (wholemeal toast) on their first study visit and on their second study visit they will be asked to eat the meal in the reverse order. The order in which this occurs will be randomised and each participant will act as their own control.
  Interventions: Other: Visit 1: Protein/fat then carbohydrate. Visit 2: Carbohydrate then protein/fat.
- Visit 1: Carbohydrate then protein/fat. Visit 2: Protein/fat then carbohydrate." (Experimental): Participants who are randomised to eat the carbohydrate-based component (wholemeal toast) of the meal before the protein/fat-based component (scrambled egg) on their first study visit and on their second study visit they will be asked to eat the meal in the reverse order. The order in which this occurs will be randomised and each participant will act as their own control.
  Interventions: Other: Visit 1: Carbohydrate then protein/fat. Visit 2: Protein/fat then carbohydrate.

INTERVENTIONS:
Other: Visit 1: Protein/fat then carbohydrate. Visit 2: Carbohydrate then protein/fat. — Participants who are randomised to eat the protein/fat-based component (scrambled egg) of the meal before the carbohydrate-based component (wholemeal toast) on their first study visit, will be asked to eat the meal in the reverse order at their second study visit. Meals will be prepared by members of the research team who have completed Food Safety training. Participants will be asked to consume a 440kcal breakfast meal within 10 minutes, approximately 1.5 hours after arrival at their first study visit and approximately 30 minutes after arrival at their second study visit.
  Arms: Visit 1: Protein/fat then carbohydrate. Visit 2: Carbohydrate then protein/fat.
Other: Visit 1: Carbohydrate then protein/fat. Visit 2: Protein/fat then carbohydrate. — Participants who are randomised to eat the carbohydrate-based component (wholemeal toast) of the meal before the protein/fat-based component (scrambled egg) on their first study visit, will be asked to eat the meal in the reverse order at their second study visit. Meals will be prepared by members of the research team who have completed Food Safety training. Participants will be asked to consume a 440kcal breakfast meal within 10 minutes, approximately 1.5 hours after arrival at their first study visit and approximately 30 minutes after arrival at their second study visit.
  Arms: Visit 1: Carbohydrate then protein/fat. Visit 2: Protein/fat then carbohydrate."

SUMMARY:
The goal of this clinical trial is to determine whether the sequence of macronutrient consumption affects post-prandial glycaemia in women with gestational diabetes mellitus.

The main questions it aims to answer are:

* The difference in the magnitude of postprandial rise in blood glucose between the two test meals.
* The difference in the magnitude of postprandial change in serum levels of gut hormones between the two test meals.
* The difference in mean change in pre-post ingestion satiety scores between the two test meals.
* The difference in 24 hour energy and macronutrient intake following the two test meals.

Participants will attend two study visits at the Centre for Public Health, with an interval of at least two days between the visits and complete the following, anthropometric measurements, demographic and appetite questionnaires, glucose measurements, two food diaries and fasting blood samples and the consumption of the study breakfast. Participants will be asked to eat either the protein/fat-based component of the meal (scrambled egg) before or after the carbohydrate-based component (wholemeal toast) on their first visit and on the other visit they will be asked to eat the meal in the reverse order. The order in which this occurs will be randomised and each participant will act as their own control. Researchers will compare the results from participants between the two test meals to see if the order of macronutrient consumption has any effect on post-prandial glycaemia, gut hormones, satiety scores and energy and macronutrient intake.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is glucose intolerance with onset or first diagnosis during pregnancy, affecting around 1 in 10 pregnancies in the United Kingdom (UK). Women with GDM are 10 times more likely to develop type 2 DM and twice as likely to develop cardiovascular disease in later life than women without GDM. Dietary modification is recommended as first line management to optimise blood glucose control. However, this often fails, necessitating the use of medication such as metformin and insulin. There is a pressing need to find safe and effective dietary approaches to optimise glycaemic control in GDM which can be easily adhered to in order to improve longer-term outcomes. The impact of the sequence of macronutrients on glycaemic control is an emerging area of interest. Recent evidence suggests that the consumption of the fat/protein components of a meal prior to the carbohydrate components, reduces the peak by around 40% after food. This study aims to determine whether the order that macronutrients (i.e. protein, fat, carbohydrate) are eaten affects; blood sugar glucose levels in the blood after a meal, appetite, food intake and the release of hormones in the body, in women with GDM.

Pregnant women with GDM, aged 18-50 years old are eligible for the study. Women are not eligible if they have a history of type 1 or 2 diabetes, any clinically confirmed food allergies, taking medication for GDM, severe nausea or using anti-sickness medication.

Recruitment will be via antenatal clinics in the South-Eastern Health and Social Care Trust (SEHSCT). Participants will attend the Centre for Public Health on two occasions (maximum 2 weeks between visits) and will involve the collection of demographic information, weight and height measurements, blood samples, glucose measurements, consumption of study breakfast, and completion of two 1-day food diaries.

Participants will be asked to eat either the protein/fat-based component of the meal (scrambled egg) before or after the carbohydrate-based component (wholemeal toast) on their first visit and on the other visit they will be asked to eat the meal in the reverse order. The order in which this occurs will be randomised and each participant will act as their own control. Scrambled egg was chosen as the protein and fat will be homogenously distributed (compared to boiled egg, for example). Wholemeal toast was chosen as, although lower glycaemic index and therefore less likely to expeditiously raise blood glucose than toasted white bread, it will be more consistent with the participants' existing dietary needs.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational diabetes mellitus
* Aged 18-50 years old

Exclusion Criteria:

* History of type 1 or type 2 diabetes mellitus
* Dietary restrictions or clinically confirmed food allergies that may affect study requirements
* Pharmacologically managed GDM at the point of study entry
* Hyperemesis gravidarum at the point of study entry (i.e. prolonged/severe nausea and vomiting)
* Using antiemetic medication (e.g. dimenhydrinate, prochlorperazine, promethazine)
* Any other problems or medical conditions that would substantially limit their ability to complete the study requirements

Participants can be recruited onto the study if they have previously had GDM in another pregnancy. Participants can also be recruited if they are involved in other research studies, but this will depend on the study type and the decision will be made by the Chief/Principal Investigator.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants must be pregnant with GDM to take part in the study, and therefore must be female.
Enrollment: 35 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial Glucose | Difference between Visit 1 [time 0 and 125 minutes] and Visit 2 [time 0 and 125 minutes]
  The difference in the magnitude of postprandial rise in blood glucose between the two test meals.

SECONDARY OUTCOMES:
Insulin | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in the magnitude of postprandial change in serum levels of insulin between the two test meals.
C-Peptide | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in the magnitude of postprandial change in serum levels of c-peptide between the two test meals.
Total Ghrelin | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in the magnitude of postprandial change in serum levels of total ghrelin between the two test meals.
Glucagon (GCG) | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in the magnitude of postprandial change in serum levels of GCG between the two test meals.
Glucagon-like peptide-1 (GLP-1) | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in the magnitude of postprandial change in serum levels of GLP-1 between the two test meals.
Peptide Tyrosine (PYY) | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in the magnitude of postprandial change in serum levels of PYY between the two test meals.
Satiety Scores | Difference between Visit 1 [time 0 and 30 minutes] and Visit 2 [time 0 and 30 minutes]
  The difference in mean change in pre-post ingestion satiety scores between the two test meals, using an appetite visual analogue scale (range 0 - 100) [The direction of the score will depend on the individual question].
Nutrient intake | Difference between Visit 1 [time 0 and 24 hours] and Visit 2 [time 0 and 24 hours]
  The difference in 24 hour energy and macronutrient intake following the two test meals.

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Centre for Public Health, Institute of Clinical Sciences A, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The researchers are happy to share results from the study for the purposes of a meta-analysis. This will be completed on approach to the researchers.
Supporting Information: Study Protocol, ICF
Time Frame: Data should be available from December 2025 and will be available for 2 years.
Access Criteria: Use of results in a meta-analysis will be available by contacting the research team.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT06896799/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT06896799/ICF_001.pdf